CLINICAL TRIAL: NCT01650311
Title: Investigating Serotonin Signalling in IBD Patients
Acronym: IBD
Status: Recruiting | Type: Observational
Sponsor: McMaster University (Other)
Responsible Party: Sponsor
Other Study IDs: 12-239
Record Dates: First submitted 2012-06-17; First posted 2012-07-26 (Estimated); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Inflammatory Bowel Disease
Keywords: IBD, CD, UC, Serotonin, 5-HT
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Samples will be collected from inflamed and non-inflamed regions, spanning the distal colon to distal ileum.
Oversight: Data Monitoring Committee: No | US Export: No

GROUPS / COHORTS (3):
- Healthy controls: Healthy control group will include participants consenting prior to colorectal cancer screening.
- CD patient groups: The patient groups will include patients with clinical diagnosis of CD.
- UC patient group: The patient groups will include patients with clinical diagnosis of UC.

SUMMARY:
Alterations in normal serotonin (5-hydroxytryptamine;5-HT) signaling have been reported in ulcerative colitis (UC) and Crohn's disease (CD). Studies report an increase in enterochromaffin (EC) cell, main source of 5-HT in the gut, numbers in CD and UC patients. Up-regulated expression of mucosal Tryptophan hydroxylase (TPH)-1, catalytic enzyme in 5-HT production, messenger RNA (mRNA) have been found in CD patients in remission who are suffering the irritable bowel syndrome (IBS)-like symptoms. Alterations in normal 5-HT signaling has also been reported in animal models of inflammatory bowel disease (IBD). Thus, the aim of the proposed research project will be to study the alterations in 5-HT signalling accompanying GI inflammatory conditions, such as IBD.

DETAILED DESCRIPTION:
The gut produces approximately 95% of serotonin (5-hydroxytryptamine; 5-HT) found in the human body; where, it is a very important mucosal signaling molecule participating in gut motility, sensation, and secretion.The vast majority of the gut-derived 5-HT is produced by specialized epithelial cells of The GI tract, called enterochromaffin (EC) cells. EC cells produce 5-HT from dietary tryptophan, this process involves the rate limiting enzyme tryptophan hydroxylase (TPH) 1, once produced this 5-HT can be released into the gut lumen, surrounding tissue and can enter the blood circulation.5-HT mediates many gastrointestinal functions, including secretion and peristalsis, by acting on a diverse range of 5-HT receptors. Five of the seven known receptor families of 5-HT (5-HT1, 5-HT2, 5-HT3, 5-HT4 and 5-HT7) are expressed in the gut.

5-HT has been evaluated in IBD and in animal models of colitis. An increase in numbers of EC cells expressing 5-HT is observed in CD and UC patients and consumption of selective 5-HT reuptake inhibitors is associated with microscopic colitis. In the present study, we plan to investigate the key elements of mucosal 5-HT signaling in CD patients for a better understanding of the role of 5-HT in pathogenesis of IBD.

ELIGIBILITY:
Inclusion Criteria:

* Patient groups: Disease diagnosis (CD or UC),duration of disease, previous/type of treatments, duration of treatment and disease prognosis.
* Healthy controls: No diagnosis of CD or UC and no diagnosis of IBS.

Exclusion Criteria:

* Patient groups: Drugs that directly affect components of 5-HT signaling, any other disease or condition that may interfere with study assessments as judged by the investigator.
* Healthy controls:Chronic use of any anti-inflammatory drugs, drugs that directly affect components of 5-HT signalling and any other disease or condition that may interfere with study assessments as judged by the investigator.

Ages: 19 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All potential participants will be included only if they meet the stringent inclusion criteria in place. Only when their eligibility is confirmed the potential participants will be approached for consent prior to endoscopy. For healthy subjects, they will be screened and consented from the colorectal screening list, also prior to endoscopy.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2012-07; Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
TPH1 | At the time of sample collection
  Levels of the gene expression and/or protein quantifications of the enzyme Tph1 will be measured to assess production of 5HT.

SECONDARY OUTCOMES:
Receptor expressions | At the time of sample collection
  Levels of the various serotonin receptors will be measured to assess changes in serotonin signaling

CONTACTS AND LOCATIONS:
Overall Officials: Waliul I Khan, MBBS, PhD., Principal Investigator — Dept. of Pathology & Molecular Medicine, McMaster University, Hamilton, Canada.; John Marshall, MD, MSc, FRCPC, AGAF., Principal Investigator — Department of Medicine, McMaster University, Hamilton, Canada.
Locations (1):
- McMaster University Medical Center, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Coates MD, Mahoney CR, Linden DR, Sampson JE, Chen J, Blaszyk H, Crowell MD, Sharkey KA, Gershon MD, Mawe GM, Moses PL. Molecular defects in mucosal serotonin content and decreased serotonin reuptake transporter in ulcerative colitis and irritable bowel syndrome. Gastroenterology. 2004 Jun;126(7):1657-64. doi: 10.1053/j.gastro.2004.03.013. PMID 15188158
- [Background] Minderhoud IM, Oldenburg B, Schipper ME, ter Linde JJ, Samsom M. Serotonin synthesis and uptake in symptomatic patients with Crohn's disease in remission. Clin Gastroenterol Hepatol. 2007 Jun;5(6):714-20. doi: 10.1016/j.cgh.2007.02.013. Epub 2007 May 4. PMID 17481962
- [Background] El-Salhy M, Danielsson A, Stenling R, Grimelius L. Colonic endocrine cells in inflammatory bowel disease. J Intern Med. 1997 Nov;242(5):413-9. doi: 10.1046/j.1365-2796.1997.00237.x. PMID 9408072
- [Background] Sharkey KA, Mawe GM. Neuroimmune and epithelial interactions in intestinal inflammation. Curr Opin Pharmacol. 2002 Dec;2(6):669-77. doi: 10.1016/s1471-4892(02)00215-1. PMID 12482729
- [Background] Khan WI, Ghia JE. Gut hormones: emerging role in immune activation and inflammation. Clin Exp Immunol. 2010 Jul 1;161(1):19-27. doi: 10.1111/j.1365-2249.2010.04150.x. Epub 2010 Apr 9. PMID 20408856
- [Background] Buchan AM. Nutrient Tasting and Signaling Mechanisms in the Gut III. Endocrine cell recognition of luminal nutrients. Am J Physiol. 1999 Dec;277(6):G1103-7. doi: 10.1152/ajpgi.1999.277.6.G1103. PMID 10600808
- [Background] Rindi G, Kloppel G. Endocrine tumors of the gut and pancreas tumor biology and classification. Neuroendocrinology. 2004;80 Suppl 1:12-5. doi: 10.1159/000080733. PMID 15477709
- [Background] Gordon JI, Schmidt GH, Roth KA. Studies of intestinal stem cells using normal, chimeric, and transgenic mice. FASEB J. 1992 Sep;6(12):3039-50. doi: 10.1096/fasebj.6.12.1521737.
- [Background] Lomax AE, Linden DR, Mawe GM, Sharkey KA. Effects of gastrointestinal inflammation on enteroendocrine cells and enteric neural reflex circuits. Auton Neurosci. 2006 Jun 30;126-127:250-7. doi: 10.1016/j.autneu.2006.02.015. Epub 2006 Apr 17. PMID 16616704
- [Background] Nagata K, Fujimiya M, Sugiura H, Uehara M. Intracellular localization of serotonin in mast cells of the colon in normal and colitis rats. Histochem J. 2001 Sep-Oct;33(9-10):559-68. doi: 10.1023/a:1014960026247. PMID 12005028
- [Background] Bertrand PP, Bertrand RL. Serotonin release and uptake in the gastrointestinal tract. Auton Neurosci. 2010 Feb 16;153(1-2):47-57. doi: 10.1016/j.autneu.2009.08.002. Epub 2009 Sep 2. PMID 19729349
- [Background] Spiller R. Serotonin and GI clinical disorders. Neuropharmacology. 2008 Nov;55(6):1072-80. doi: 10.1016/j.neuropharm.2008.07.016. Epub 2008 Jul 19. PMID 18687345
- [Background] Belai A, Boulos PB, Robson T, Burnstock G. Neurochemical coding in the small intestine of patients with Crohn's disease. Gut. 1997 Jun;40(6):767-74. doi: 10.1136/gut.40.6.767. PMID 9245931
- [Background] Wheatcroft J, Wakelin D, Smith A, Mahoney CR, Mawe G, Spiller R. Enterochromaffin cell hyperplasia and decreased serotonin transporter in a mouse model of postinfectious bowel dysfunction. Neurogastroenterol Motil. 2005 Dec;17(6):863-70. doi: 10.1111/j.1365-2982.2005.00719.x. PMID 16336502
- [Background] Gershon MD. Serotonin and its implication for the management of irritable bowel syndrome. Rev Gastroenterol Disord. 2003;3 Suppl 2:S25-34. PMID 12776000
- [Background] Kim DY, Camilleri M. Serotonin: a mediator of the brain-gut connection. Am J Gastroenterol. 2000 Oct;95(10):2698-709. doi: 10.1111/j.1572-0241.2000.03177.x. No abstract available. PMID 11051338
- [Background] Oshima S, Fujimura M, Fukimiya M. Changes in number of serotonin-containing cells and serotonin levels in the intestinal mucosa of rats with colitis induced by dextran sodium sulfate. Histochem Cell Biol. 1999 Oct;112(4):257-63. doi: 10.1007/s004180050445. PMID 10550609
- [Background] Linden DR, Chen JX, Gershon MD, Sharkey KA, Mawe GM. Serotonin availability is increased in mucosa of guinea pigs with TNBS-induced colitis. Am J Physiol Gastrointest Liver Physiol. 2003 Jul;285(1):G207-16. doi: 10.1152/ajpgi.00488.2002. Epub 2003 Mar 19. PMID 12646422
- [Background] Yang GB, Lackner AA. Proximity between 5-HT secreting enteroendocrine cells and lymphocytes in the gut mucosa of rhesus macaques (Macaca mulatta) is suggestive of a role for enterochromaffin cell 5-HT in mucosal immunity. J Neuroimmunol. 2004 Jan;146(1-2):46-9. doi: 10.1016/j.jneuroim.2003.10.044. PMID 14698846
- [Background] Wang H, Steeds J, Motomura Y, Deng Y, Verma-Gandhu M, El-Sharkawy RT, McLaughlin JT, Grencis RK, Khan WI. CD4+ T cell-mediated immunological control of enterochromaffin cell hyperplasia and 5-hydroxytryptamine production in enteric infection. Gut. 2007 Jul;56(7):949-57. doi: 10.1136/gut.2006.103226. Epub 2007 Feb 15. PMID 17303597
- [Background] Spiller R. Serotonin, inflammation, and IBS: fitting the jigsaw together? J Pediatr Gastroenterol Nutr. 2007 Dec;45 Suppl 2:S115-9. doi: 10.1097/MPG.0b013e31812e66da. PMID 18185071
- [Background] Gershon MD, Tack J. The serotonin signaling system: from basic understanding to drug development for functional GI disorders. Gastroenterology. 2007 Jan;132(1):397-414. doi: 10.1053/j.gastro.2006.11.002. PMID 17241888
- [Background] Idzko M, Panther E, Stratz C, Muller T, Bayer H, Zissel G, Durk T, Sorichter S, Di Virgilio F, Geissler M, Fiebich B, Herouy Y, Elsner P, Norgauer J, Ferrari D. The serotoninergic receptors of human dendritic cells: identification and coupling to cytokine release. J Immunol. 2004 May 15;172(10):6011-9. doi: 10.4049/jimmunol.172.10.6011. PMID 15128784
- [Background] Leon-Ponte M, Ahern GP, O'Connell PJ. Serotonin provides an accessory signal to enhance T-cell activation by signaling through the 5-HT7 receptor. Blood. 2007 Apr 15;109(8):3139-46. doi: 10.1182/blood-2006-10-052787. Epub 2006 Dec 7. PMID 17158224
- [Background] Meredith EJ, Chamba A, Holder MJ, Barnes NM, Gordon J. Close encounters of the monoamine kind: immune cells betray their nervous disposition. Immunology. 2005 Jul;115(3):289-95. doi: 10.1111/j.1365-2567.2005.02166.x. PMID 15946246
- [Background] Young MR, Matthews JP. Serotonin regulation of T-cell subpopulations and of macrophage accessory function. Immunology. 1995 Jan;84(1):148-52. PMID 7890297
- [Background] Ghia JE, Li N, Wang H, Collins M, Deng Y, El-Sharkawy RT, Cote F, Mallet J, Khan WI. Serotonin has a key role in pathogenesis of experimental colitis. Gastroenterology. 2009 Nov;137(5):1649-60. doi: 10.1053/j.gastro.2009.08.041. Epub 2009 Aug 23. PMID 19706294
- [Background] Wirtz S, Neufert C, Weigmann B, Neurath MF. Chemically induced mouse models of intestinal inflammation. Nat Protoc. 2007;2(3):541-6. doi: 10.1038/nprot.2007.41. PMID 17406617
- [Background] Costedio MM, Hyman N, Mawe GM. Serotonin and its role in colonic function and in gastrointestinal disorders. Dis Colon Rectum. 2007 Mar;50(3):376-88. doi: 10.1007/s10350-006-0763-3. PMID 17195902
- [Background] Heller F, Florian P, Bojarski C, Richter J, Christ M, Hillenbrand B, Mankertz J, Gitter AH, Burgel N, Fromm M, Zeitz M, Fuss I, Strober W, Schulzke JD. Interleukin-13 is the key effector Th2 cytokine in ulcerative colitis that affects epithelial tight junctions, apoptosis, and cell restitution. Gastroenterology. 2005 Aug;129(2):550-64. doi: 10.1016/j.gastro.2005.05.002. PMID 16083712
- [Background] Kidd M, Gustafsson BI, Drozdov I, Modlin IM. IL1beta- and LPS-induced serotonin secretion is increased in EC cells derived from Crohn's disease. Neurogastroenterol Motil. 2009 Apr;21(4):439-50. doi: 10.1111/j.1365-2982.2008.01210.x. Epub 2008 Oct 25. PMID 19019013
- [Background] Bishop AE, Pietroletti R, Taat CW, Brummelkamp WH, Polak JM. Increased populations of endocrine cells in Crohn's ileitis. Virchows Arch A Pathol Anat Histopathol. 1987;410(5):391-6. doi: 10.1007/BF00712758. PMID 3103321
- [Background] Khan WI, Motomura Y, Wang H, El-Sharkawy RT, Verdu EF, Verma-Gandhu M, Rollins BJ, Collins SM. Critical role of MCP-1 in the pathogenesis of experimental colitis in the context of immune and enterochromaffin cells. Am J Physiol Gastrointest Liver Physiol. 2006 Nov;291(5):G803-11. doi: 10.1152/ajpgi.00069.2006. Epub 2006 May 25. PMID 16728728
- [Background] Nakajima M, Shiihara Y, Shiba Y, Sano I, Sakai T, Mizumoto A, Itoh Z. Effect of 5-hydroxytryptamine on gastrointestinal motility in conscious guinea-pigs. Neurogastroenterol Motil. 1997 Dec;9(4):205-14. doi: 10.1046/j.1365-2982.1997.d01-56.x. PMID 9430788
- [Background] Li N, Ghia JE, Wang H, McClemens J, Cote F, Suehiro Y, Mallet J, Khan WI. Serotonin activates dendritic cell function in the context of gut inflammation. Am J Pathol. 2011 Feb;178(2):662-71. doi: 10.1016/j.ajpath.2010.10.028. PMID 21281798
- [Background] Magro F, Vieira-Coelho MA, Fraga S, Serrao MP, Veloso FT, Ribeiro T, Soares-da-Silva P. Impaired synthesis or cellular storage of norepinephrine, dopamine, and 5-hydroxytryptamine in human inflammatory bowel disease. Dig Dis Sci. 2002 Jan;47(1):216-24. doi: 10.1023/a:1013256629600. PMID 11837726
- [Background] Wong JM, Wei SC. Efficacy of Pentasa tablets for the treatment of inflammatory bowel disease. J Formos Med Assoc. 2003 Sep;102(9):613-9. PMID 14625605
- [Background] Cremon C, Carini G, Wang B, Vasina V, Cogliandro RF, De Giorgio R, Stanghellini V, Grundy D, Tonini M, De Ponti F, Corinaldesi R, Barbara G. Intestinal serotonin release, sensory neuron activation, and abdominal pain in irritable bowel syndrome. Am J Gastroenterol. 2011 Jul;106(7):1290-8. doi: 10.1038/ajg.2011.86. Epub 2011 Mar 22. PMID 21427712